CLINICAL TRIAL: NCT07289919
Title: Exploring Sustainable Alternatives to Marine Oils: A Clinical Trial on the Efficacy of Echium and Ahiflower Oils for Omega-3 Supplementation.
Brief Title: Exploring Sustainable Alternatives to Marine Oils With Echium and Ahiflower Oils
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Inar Castro Erger, Full Professor, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 85126524.0.0000.0067
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular (CV) Risk; Atheroscleroses; Inflamation; Omega 3 Fatty Acids; Supplement
Keywords: Omega - 3 fatty acids; stearidonic acid; fish oil; Echium oil; Ahiflower oil; Humans; Crossover
MeSH Terms: conditions — Atherosclerosis | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Crossover Intervention Sequence 1 (Experimental): All participants will receive all three interventions (Echium oil, Ahiflower® oil, and EPA capsules) in a randomized crossover sequence. Each intervention period lasts 8 weeks, followed by a 4-week washout period. Participants rotate through all treatments, ensuring within-subject comparison. In this sequence, participants begin with Echium oil, transition to EPA capsules, and complete the cycle with Ahiflower oil.
  Interventions: Dietary Supplement: Echium oil; Dietary Supplement: Ahiflower oil; Dietary Supplement: EPA capsules
- Crossover Intervention Sequence 2 (Experimental): All participants will receive all three interventions (Echium oil, Ahiflower® oil, and EPA capsules) in a randomized crossover sequence. Each intervention period lasts 8 weeks, followed by a 4-week washout period. Participants rotate through all treatments, ensuring within-subject comparison. In this sequence, participants begin with Ahiflower oil, transition to Echium oil, and complete the cycle with EPA capsules.
  Interventions: Dietary Supplement: Echium oil; Dietary Supplement: Ahiflower oil; Dietary Supplement: EPA capsules
- Crossover Intervention Sequence 3 (Experimental): All participants will receive all three interventions (Echium oil, Ahiflower® oil, and EPA capsules) in a randomized crossover sequence. Each intervention period lasts 8 weeks, followed by a 4-week washout period. Participants rotate through all treatments, ensuring within-subject comparison. In this sequence, participants begin with EPA capsules, transition to Ahiflower oil, and complete the cycle with Echium oil.
  Interventions: Dietary Supplement: Echium oil; Dietary Supplement: Ahiflower oil; Dietary Supplement: EPA capsules

INTERVENTIONS:
Dietary Supplement: Echium oil — Participants consume 15 g/day of Echium oil, incorporated into meals, during one 8-week phase.
  Other Names: seed oil from Echium plantagineum
Dietary Supplement: Ahiflower oil — Participants consume 15 g/day of Ahiflower® oil, incorporated into meals, during one 8-week phase.
  Other Names: Buglossoides arvensis; Lithospermum arvense; corn gromwell
Dietary Supplement: EPA capsules — Participants consume three EPA capsules daily (totaling 2.34 g/day), taken with meals, during one 8-week phase.
  Other Names: Omega-3; IPE

SUMMARY:
This randomized, single-blind, crossover clinical trial aims to evaluate Echium oil and Ahiflower® oil as sustainable, plant-based alternatives to marine oils for omega-3 supplementation. Although fish oil is the primary dietary source of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), its use as a dietary supplementation presents several drawbacks, including high cost, potential contamination, limited global supply, and sustainability concerns. Echium and Ahiflower oils are naturally rich in stearidonic acid (SDA), a metabolic intermediate that bypasses the rate-limiting Δ6-desaturase step in the omega-3 pathway, potentially enhancing the conversion to EPA.

Fifteen participants will undergo three 8-week intervention phases-Echium oil (15 g/day), Ahiflower oil (15 g/day), or EPA capsules (2.34 g/day)-separated by four-week washout periods. Blood samples will be collected before and after each phase to measure fatty acid profiles in plasma, plasma fractions, and erythrocytes using GC-MS. Anthropometric and biochemical parameters will also be assessed. The study seeks to determine whether SDA-rich plant oils can effectively increase EPA levels in humans and potentially reduce the reliance on marine oils for cardiovascular health benefits.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will include individuals of both sexes, aged 18 to 30 years, without contraindications for using fish oil or vegetable oil supplements. Women must not be pregnant or breastfeeding.

Exclusion Criteria:

* will include vegetarianism or veganism; the use of triglyceride-lowering medications or dietary supplements; consumption of fish oil or other n-3 or n-6 PUFA supplements/drugs within one month before the trial; consumption of fatty fish (salmon, herring, mackerel, albacore tuna, or sardines) more than twice a month in the month before the trial; and unwillingness to avoid PUFA supplements and seafood throughout the study period. Additional exclusions will include severe heart failure, active severe liver disease, planned coronary intervention or surgery, history of acute or chronic pancreatitis, known hypersensitivity to fish, shellfish, or capsule ingredients, and autoimmune diseases requiring immunosuppressive therapy or current systemic corticosteroid use. Other exclusion criteria will encompass active neoplasms requiring surgery, chemotherapy, or radiation within the past 12 months (patients who underwent curative surgery without further treatment in the last 12 months may be eligible); inflammatory bowel disease or chronic diarrhea; significant non-transient hematological abnormalities; renal dysfunction; severe liver disease; inability to provide informed consent; participation in another clinical trial involving an investigational agent within the past 90 days; malabsorption syndrome; recent drug or alcohol abuse; atrial fibrillation; or bleeding disorders. Adherence to the prescribed dosage will be assessed by tracking the residual oil sachets and capsules returned by participants. If fewer than 80% of the doses over the full study period are consumed, participants will be classified as non-compliant, and their data will be excluded from efficacy analyses.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2025-05-26 (Actual); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in EPA and DHA concentrations in blood fractions | Baseline and after each 8-week intervention phase
  EPA (eicosapentaenoic acid) and DHA (docosahexaenoic acid) concentrations will be determined from blood fractions (plasma, plasma subfractions, and erythrocytes). Lipids will be extracted and derivatized to obtain fatty acid methyl esters (FAMEs), which will then be analyzed by gas chromatography-mass spectrometry (GC-MS). Measurements will be performed at baseline and after each 8-week intervention phase (Echium oil, Ahiflower® oil, and EPA capsules) to assess the efficiency of omega-3 conversion and incorporation under each supplementation condition

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmaceutical Sciences, University of São Paulo (USP), São Paulo, São Paulo, Brazil